CLINICAL TRIAL: NCT01480674
Title: A Retrospective Study to Characterize Patients With HER2-positive Metastatic or Locally Advanced Breast Cancer, Treated by Herceptin® as 1st Line-therapy and Without Progression for at Least 3 Years Followed by a 1-year Prospective Study for Patients Still Alive
Brief Title: An Observational Study of Patients With HER2-Positive Metastatic or Locally Advanced Breast Cancer Treated With Herceptin (Trastuzumab) in 1st Line and Without Progression For 3 Years
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML23001
Record Dates: First submitted 2011-08-18; First posted 2011-11-29 (Estimated); Results first posted 2016-02-24 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2017-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

GROUPS / COHORTS (1):
- Trastuzumab: Eligible participants with human epidermal growth factor receptor 2 (HER2)-positive metastatic or locally advanced breast cancer, who were treated with trastuzumab as a first-line therapy and were progression-free for at least 3 years after treatment initiation, were included and were followed for one year.
  Interventions: Drug: Trastuzumab

INTERVENTIONS:
Drug: Trastuzumab

SUMMARY:
This observational study will characterize retrospectively patients with HER2-positive metastatic or locally advanced breast cancer who had received treatment with Herceptin (trastuzumab) in 1st line and who were without progression for at least three years. Patients will be followed prospectively for one year.

ELIGIBILITY:
Inclusion Criteria:

* Female patients, >/= 18 years of age
* HER2-positive metastatic breast cancer or locally advanced breast cancer
* Systemic treatment included Herceptin as 1st line therapy
* Without progression for at least 3 years after the beginning of Herceptin treatment
* Alive or not alive and treated or not treated with Herceptin at the time of inclusion

Exclusion Criteria:

* Disease progression <3 years after beginning 1st-line therapy with Herceptin

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HER2-positive metastatic breast cancer or locally advanced breast cancer whose systemic treatment included Herceptin as 1st line therapy, and who were without progression for at least 3 years after beginning Herceptin
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2011-03-28 (Actual); Primary Completion 2012-11-16 (Actual); Study Completion 2012-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (78):
- France (78):
  - Clinique Du Docteur Calabet; Cromg, Agen
  - C.H. Du Pays D'aix En Provence Service du Dr Blanc, Aix-en-Provence
  - Poly Parc Rambot La Provencale; Chimiotherapie Ambulatoire, Aix-en-Provence
  - Chd Castelluccio; Oncologie, Ajaccio
  - Clinique De L Europe; Pmsi, Amiens
  - Clinique De L Europe; Radiotherapie Chimiotherapie, Amiens
  - HOP Prive Arras Les Bonnettes; Chimiotherapie, Arras
  - Hopital Europeen La Roseraie;Radiotherapie, Aubervilliers
  - Polyclinique Sainte Marguerite; Chimiotherapie, Auxerre
  - Clinique Champeau Mediterranee; Radiotherapie Oncologie, Béziers
  - Hopital Saint Andre; Oncologie 2, Bordeaux
  - Polyclinique Bordeaux Nord Aquitaine; Chimiotherapie Radiotherapie, Bordeaux
  - Centre Hospitalier Fleyriat; Oncologie/Hematologie, Bourg-en-Bresse
  - Hopital Augustin Morvan; Hopital De Jour, Brest
  - Ch De Brive La Gaillarde; Radiotherapie Oncologie, Brive-la-Gaillarde
  - Centre Francois Baclesse; Comite Sein, Caen
  - Ch Antoine Gayraud; Oncologie, Carcassonne
  - Clinique Montreal; Chimiotherapie, Carcassonne
  - Ch William Morey; Medecine 1, Chalon-sur-Saône
  - Centre Jean Perrin; Hopital De Jour, Clermont-Ferrand
  - Pole Sante Republique;Oncologie Hematologie, Clermont-Ferrand
  - Ch De Dax; Radiotherapie Oncologie, Dax
  - Centre Leonard De Vinci;Chimiotherapie, Dechy
  - Centre Georges Francois Leclerc; Oncologie 3, Dijon
  - Hopital Prive Drome Ardeche; Chir 2A 2B, Guilherand-Granges
  - Clinique de L' Esperance; Oncologie, Hyères
  - Polyclinique de Blois; Chimiotherapie Ambulatoire, La Chaussée-Saint-Victor
  - CH Dptal Les Oudairies; Hematologie Oncologie, La Roche-sur-Yon
  - Hopital Albert Michallon; Oncologie, La Tronche
  - Polyclinique Du Bois; Centre Bourgogne, Lille
  - Polyclinique Du Bois; Oncologie, Lille
  - Ch De Longjumeau; Hopital De Jour Et Semaine, Longjumeau
  - Clinique Des 4 Pavillons; Chimiotherapie, Lormont
  - Centre Leon Berard; Departement Oncologie Medicale, Lyon
  - Polyclinique Du Beaujolais; Chimiotherapie, Lyon
  - Hopital Edouard Herriot; Pavillon F Rhumatologie, Lyon
  - Hôpital Saint Joseph; Oncologie Medicale, Marseille
  - Polyclinique Du Val De Saone; Chimiotherapie, Mâcon
  - Ch De Montelimar; Radiotherapie, Montélimar
  - Clinique Clementville; Hopital De Jour, Montpellier
  - Polyclinique Saint Roch; Hop Jour Chimio Radiotherapie, Montpellier
  - Centre Azureen De Cancerologie; Cons externes, Mougins
  - Hopital Emile Muller; Oncologie Radiotherapie, Mulhouse
  - Centre D'Oncologie de Gentilly; Oncology, Nancy
  - Polyclinique Gentilly; CHIMIOTHERAPIE AMBULATOIRE, Nancy
  - Clinique Des Genets; Radiotherapie, Narbonne
  - Clinique Henry Hartmann; Oncologie, Neuilly-sur-Seine
  - Centre Antoine Lacassagne; Hopital De Jour A2, Nice
  - Centre Hospitalier Uni Ire Caremeau; Radiotherapie & Oncologie, Nîmes
  - Polyclinique Kenval ; Radiotherapie Oncologie, Nîmes
  - Clinique sainte marie; chimiotherapie ambulatoire, Osny
  - Hopital Saint Louis; Oncologie Medicale, Paris
  - Hopital Des Diaconesses; Hopital De Jour, Paris
  - Ch Pitie Salpetriere; Oncologie Medicale, Paris
  - HOPITAL TENON; Cancerologie Medicale, Paris
  - Clinique Francheville; Radiotherapie, Périgueux
  - Ch Lyon Sud; Hemato Secteur Jules Courmont, Pierre-Bénite
  - Ch Lyon Sud; Onco Secteur Jules Courmont, Pierre-Bénite
  - Ch De Pithiviers; Consult Externes, Pithiviers
  - Institut Jean Godinot; Pavillon Rubis, Reims
  - Polyclinique De Courlancy; Chimiotherapie Ambulatoire, Reims
  - Centre Eugene Marquis; Unite Huguenin, Rennes
  - Clinique Saint Hilaire; Sce Chimiotherapie, Rouen
  - Chp Saint Gregoire; Cancerologie Radiotherapie, Saint-Grégoire
  - Ico Rene Gauducheau; Oncologie, Saint-Herblain
  - Clinique de L'Union; Oncologie, Saint-Jean
  - Centre Radiotherapie Etienne Dolet, Saint-Nazaire
  - Institut De Cancerologie De La Loire; Consult Oncologie Niveau 0, Saint-Priest-en-Jarez
  - Ch De Saint Quentin; Medecine B10, Saint-Quentin
  - CH De Senlis; Medecine 2, Senlis
  - Ch De Soissons; Medecine Ambulatoire, Soissons
  - Institut Claudius Regaud; Departement Oncologie Medicale, Toulouse
  - Clinique Pasteur; Oncologie Medicale, Toulouse
  - Chevelle Christian; Centre De Radiotherapie, Toulouse
  - Centre Alexis Vautrin; Oncologie Medicale, Vandœuvre-lès-Nancy
  - Hopital Saint Nicolas; Pneumologie, Verdun
  - Institut Gustave Roussy; Comite 5, Villejuif
  - Institut Gustave Roussy; Departement Oncologie Medicale, Villejuif

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 160 participants were recruited from 28 March 2011 to 16 November 2012.
Groups:
- Trastuzumab: Eligible participants with human epidermal growth factor receptor 2 (HER2)-positive metastatic or locally advanced breast cancer, who were treated with trastuzumab (Herceptin) as a first-line therapy and were progression-free for at least 3 years after treatment initiation, were included and were followed for one year.
Period: Overall Study
Arm/Group | Trastuzumab
Started | 160
Safety Set | 154
Analysed Set | 128
Completed | 125
Not Completed | 35
Not completed — Death | 23
Not completed — Lost to Follow-up | 2
Not completed — visit not done | 10

BASELINE CHARACTERISTICS:
Population: Analyzed set population included all enrolled participants without any protocol deviation used as a primary analysis population for all efficacy outcome measures.
Groups:
- Trastuzumab: Eligible participants with HER2-positive metastatic or locally advanced breast cancer, who were treated with trastuzumab as a first-line therapy and were progression-free for at least 3 years after treatment initiation, were included and were followed for one year.
Arm/Group | Trastuzumab
Number analyzed (Participants) | 128
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.3 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Tumor Hormone Receptor Status of Participants Without Progression
Description: The clinical and tumor characteristics including HER2 and Hormone Receptor (HR) status of metastatic breast cancer participants are analysed which are important factors which impact on Progression Free Survival.
Time Frame: Up to 3 years
Population: Analyzed set population included all enrolled participants without any protocol deviation. This population set was used as a primary analysis population for all efficacy outcome measures. Participants with available data at the time of evaluation were reported.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Trastuzumab
Number analyzed (Participants) | 125
Percentage of participants
  HR Positive | 57.6 [48.8 to 65.9]
  HR Negative | 42.4 [34.1 to 51.2]

2. Primary Outcome: Percentage of Participants With Prevalence of Bone Metastases Without Progression for at Least 3 Years After the Beginning of 1st Line Herceptin Treatment
Description: Bone metastasis occurs when cancer cells spread from their original site to a bone. Percentage of participants with prevalence of bone metastases without progression were reported
Time Frame: Up to 3 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Trastuzumab
Number analyzed (Participants) | 127
Percentage of participants | 42.5 [34.3 to 51.2]

3. Secondary Outcome: Progression-free Survival
Description: The Progression-free survival (PFS) was defined as the time between the treatment start date (date of first trastuzumab infusion during the metastatic period) and the date of the first progressive disease or death from any cause. The method of assessment of disease progression was not outlined within the protocol, this was completed by each investigator in line with routine practice.
Time Frame: Up to 12 years
Population: Analyzed set population included all enrolled participants without any protocol deviation. This population set was used as a primary analysis population for all efficacy outcome measures.
Measure: Median (95% Confidence Interval); unit: Years
Arm/Group | Trastuzumab
Number analyzed (Participants) | 128
Years | 6.44 [5.68 to NA] — The value was not evaluated.

4. Secondary Outcome: Time to Progression
Description: The Time to progression (TTP) was defined as the time between the treatment start date (date of the first trastuzumab infusion during the metastatic period) and the date of the first progressive disease.
Time Frame: Up to 12 years
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Years
Arm/Group | Trastuzumab
Number analyzed (Participants) | 128
Years | 6.44 [5.77 to NA] — The value was not evaluated.

5. Secondary Outcome: Overall Survival
Description: The overall survival (OS) was defined as the time between the treatment start date (date of the first trastuzumab infusion during the metastatic period) and the death from any cause.
Time Frame: Up to 12 years
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Years
Arm/Group | Trastuzumab
Number analyzed (Participants) | 128
Years | NA [NA to NA] — Median OS not achieved (only 12.5% of participants died).

6. Secondary Outcome: Dosage Schedule of Herceptin Treatment
Description: Participants who received trastuzumab are reported in the below table. The regimen of trastuzumab in first line treatment is presented as in frequency 1 infusion (inf) per week (W) and dose per infusion as mg/kg.
Time Frame: Up to 12 years
Population: Analyzed set population included all enrolled participants without any protocol deviation. This population set was used as a primary analysis population for all efficacy outcome measures. Participants with available data at specified time points are denoted as 'n'.
Measure: Number; unit: Participants
Arm/Group | Trastuzumab
Number analyzed (Participants) | 125
Participants
  Dose and frequency of inf:1 inf / W, n= 125 | 40
  1 inf/2W, n= 125 | 2
  1 inf / 3W, n= 125 | 82
  3 inf/4W, n= 125 | 1
  Dose per inf: 2 mg/kg, n= 124 | 10
  3 mg/kg, n= 124 | 1
  4 mg/kg, n= 124 | 39
  6 mg/kg, n= 124 | 25
  8 mg/kg, n= 124 | 49

7. Secondary Outcome: Number of Participants With Antineoplastic Treatment in Combination With Trastuzumab and After Discontinuation of Trastuzumab Treatment
Description: Antineoplastic treatment given in combination with and after discontinuation (Aft. Dis) of herceptin treatment included chemotherapy and hormonotherapy.
Time Frame: Up to 12 years
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | Trastuzumab
Number analyzed (Participants) | 128
Participants
  With Trastuzumab, Chemotherapy, n= 119 | 117
  With Trastuzumab, Hormonotherapy, n= 51 | 50
  Aft. Dis, Chemotherapy n= 128 | 22
  Aft. Dis, hormonotherapy n= 128 | 4

8. Secondary Outcome: Number of Participants With Any Adverse Events and Serious Adverse Events
Description: An adverse event (AE) was defined as any untoward medical occurrence that occurred during the course of the trial after study treatment had started. An adverse event was therefore any unfavourable and unintended sign, symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. A Serious Adverse Event (SAE) is any untoward medical occurrence that at any dose results in death, are life threatening, requires hospitalization or prolongation of hospitalization or results in disability/incapacity, and congenital anomaly/birth defect. The data was reported for prospective period.
Time Frame: Up to 1 year
Population: The safety population set included of all participants who received at least one dose of study drug. Participants with available data in the prospective period were analysed.
Measure: Number; unit: Participants
Arm/Group | Trastuzumab
Number analyzed (Participants) | 134
Participants
  Any AEs | 30
  Any SAEs | 6

9. Secondary Outcome: The Duration of Treatment of Trastuzumab
Description: Total treatment duration and duration of the first line of treatment is reported.
Time Frame: Up to 1 Year
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | Trastuzumab
Number analyzed (Participants) | 128
Years
  First line of treatment | 4.89 (2.13)
  Total treatment duration | 5.57 (2.36)

ADVERSE EVENTS:
Time Frame: Up to 1 year
Description: An AE is defined as any unfavourable and unintended sign, symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug .The data was reported for prospective period. Participants with available data in the prospective period were analysed.
Arm/Group | Trastuzumab
Serious Adverse Events (participants affected / at risk) | 6/134
Other Adverse Events (participants affected / at risk) | 30/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab (N=134)
Paraplegia (Nervous system disorders) | 1
Coma (Nervous system disorders) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Lymphoedema (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab (N=134)
Leukopenia (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 1
Atrioventricular extrasystoles (Cardiac disorders) | 1
Left ventricular dysfunction (Cardiac disorders) | 1
Deafness (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 3
Cushing's syndrome (Endocrine disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Aphthous stomatitis (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 5
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2
Gingival bleeding (Gastrointestinal disorders) | 1
Gingivitis (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 3
Rectal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 6
Chest discomfort (General disorders) | 1
Chest pain (General disorders) | 1
Fatigue (General disorders) | 1
Mucosal inflammation (General disorders) | 1
Oedema (General disorders) | 1
Oedema peripheral (General disorders) | 2
Cytolytic hepatitis (Hepatobiliary disorders) | 1
Erysipelas (Infections and infestations) | 1
Herpes virus infection (Infections and infestations) | 1
Sinobronchitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 3
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1
Radiation skin injury (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Blood glucose (Investigations) | 1
Blood sodium (Investigations) | 1
Ejection fraction decreased (Investigations) | 1
Gamma-glutamyltransferase (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hypercreatininaemia (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 1
Brain oedema (Nervous system disorders) | 1
Headache (Nervous system disorders) | 3
Neuropathy peripheral (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Paresis (Nervous system disorders) | 1
Sciatic nerve neuropathy (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 4
Rosacea (Skin and subcutaneous tissue disorders) | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 2
Cataract operation (Surgical and medical procedures) | 1
Mastectomy (Surgical and medical procedures) | 1
Ischaemic limb pain (Vascular disorders) | 1
Lymphoedema (Vascular disorders) | 2
Subclavian vein thrombosis (Vascular disorders) | 1
Thrombophlebitis superficial (Vascular disorders) | 1
Vascular compression (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.